CLINICAL TRIAL: NCT03148418
Title: An Open-Label, Multicenter Extension and Long-Term Observational Study in Patients Previously Enrolled in a Genentech- and/or F. Hoffmann-La Roche Ltd-Sponsored Atezolizumab Study
Brief Title: A Study in Participants Previously Enrolled in a Genentech- and/or F. Hoffmann-La Roche Ltd-Sponsored Atezolizumab Study (IMbrella A)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO39633; 2016-005189-75 (EudraCT Number)
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Atezolizumab Monotherapy (Experimental): Participants will continue to receive atezolizumab monotherapy in a Genentech or Roche-sponsored study (the parent study) in accordance with local prescribing information till the participant continues to derive clinical benefit or until death, withdrawal of study consent, unacceptable toxicity, pregnancy, participant non-compliance, or study termination by the Sponsor, whichever occurs first.
  Interventions: Drug: Atezolizumab
- Combined Agents with Atezolizumab (Experimental): Participants will receive treatment of atezolizumab with combined agent(s) as directed per the parent study. Participants will receive agent(s) in combination with atezolizumab at the same dose and schedule, and with the same administration guidelines that were in effect at the time of participant discontinuation from the parent study.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- Comparator Treatment (Active Comparator): Participants will receive comparator treatment administration as directed per the parent study. Participants will receive comparator treatment at the same dose and schedule, and with the same administration guidelines that were in effect at the time of participant discontinuation from the parent study.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered as a monotherapy or atezolizumab with other agent(s) as per parent protocol. Dosing regimen will continue in accordance with the parent study or at equivalent dose (if applicable) and at the same schedule as the parent study, or switch to a fixed atezolizumab dose of 1200 mg every 3 weeks (Q3W).
  Other Names: RO5541267; Tecentriq
  Arms: Atezolizumab Monotherapy; Combined Agents with Atezolizumab
Drug: Bevacizumab — Bevacizumab will be administered as directed per the parent study.
  Other Names: Avastin
  Arms: Combined Agents with Atezolizumab; Comparator Treatment

SUMMARY:
This is an open-label, multicenter, non-randomized extension and long-term observational study. Participants receiving atezolizumab monotherapy or atezolizumab combined with other agent(s) or comparator agent(s) in a Genentech or Roche-sponsored study (the parent study) and who continue to receive study treatment at the time of the parent-study closure and do not have access to the study treatment locally are eligible for continued treatment in the extension study. Dosing regimen for a given participant and indication will be the same or equivalent to the respective parent study protocol. Study treatment in the extension study can continue until disease progression or beyond if the patient continues to derive clinical benefit as judged by the investigator and if allowed by the parent study or local prescribing information until death; withdrawal of study consent; unacceptable toxicity; pregnancy; patient non-compliance; or study termination by the Sponsor, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

Specific criteria for patients who continue treatment as well as safety and survival follow-up in the extension study (and survival follow up for pattients who roll over from IMpower133):

* Eligible for continuing or crossing over to atezolizumab-based therapy at the time of the parent-study closure as per the parent study or eligible for continuing the comparator agent(s) in a Genentech- or Roche-sponsored study at the time of the parent-study closure as per the parent study, with no access to commercially available comparator agent
* First dose of study treatment in the extension study will be received within 7 days of the treatment interruption window allowed by the parent study
* Continue to benefit from atezolizumab-based study treatment or from the comparator at the time of parent-study closure as assessed by the investigator
* Negative serum pregnancy test within 7 days prior to start of study treatment in women of childbearing potential

Specific criteria for patients from the IMpower133 parent study only who do not continue treatment in the extension study and/or receive commercially available atezolizumab (Tecentriq) outside this extension study and continue safety and survival follow-up only in the extension study:

- Discontinuation of atezolizumab-based therapy in the IMpower133 parent study and in survival follow- up at the time of IMpower133 parent study closure, or eligible for continuing or crossing over to atezolizumab-based therapy as per the IMpower133 parent protocol and have access to commercially available atezolizumab (Tecentriq) outside this extension study at the time of the IMpower133 parent-study closure

Exclusion Criteria:

Specific criteria for patients who continue treatment as well as safety and survival follow-up in the extension study:

* Meet of any of the study treatment discontinuation criteria specified in the parent study at the time of enrollment in the extension study
* Study treatment is commercially marketed in the patient's country for the patient specific disease and is accessible to the patient
* Time between the last dose of treatment received in parent study and first dose in extension study is longer than the interruption period (± 7 days) allowed in the parent study
* Treatment with any anti-cancer treatment (other than treatment permitted in the parent study) during the time between last treatment in the parent study and the first dose of study treatment in the extension study
* Permanent discontinuation of atezolizumab for any reason during the parent study or during the time between last treatment in the parent study and the first dose of study treatment in the extension study (if applicable)
* Any unresolved or irreversible toxicities during the parent study that required permanent discontinuation of study treatment, in accordance to the parent study or local prescribing information
* Ongoing SAE(s) that has not resolved to baseline level or Grade less than or equal to (<=) 1 from the parent study or during the time between last treatment in the parent study and the first dose of study treatment in the extension study
* Any serious uncontrolled concomitant disease that would contraindicate the use of study treatment at the time of the extension study or that would place the participant at high risk for treatment-related complications
* Concurrent participation in any therapeutic clinical trial (other than the parent study)

Specific criteria for patients who do not continue treatment in the extension study and/or receive commercially available atezolizumab (Tecentriq) outside this extension study and continue safety and survival follow-up only in the extension study:

- Discontinuation of comparator in parent study and in survival follow-up at the time of parent study closure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2030-03-06 (Estimated); Study Completion 2030-03-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Continued Access to Atezolizumab-Based Therapy and/or Comparator Agent(s) | Day 1 up to maximum 10 years

SECONDARY OUTCOMES:
Percentage of Participants With Serious Adverse Events (SAEs) by Severity Determined According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 | Day 1 up to 90 days after last dose of study treatment (last dose=till clinical benefit or until death, withdrawal of consent, unacceptable toxicity, pregnancy, non-compliance, or termination by Sponsor, whichever occurs first) (up to maximum 10 years)
Percentage of Participants With Adverse Events of Special Interest by Severity Determined According to NCI CTCAE Version 4.0 | Day 1 up to 90 days after last dose of study treatment (last dose=till clinical benefit or until death, withdrawal of consent, unacceptable toxicity, pregnancy, non-compliance, or termination by Sponsor, whichever occurs first) (up to maximum 10 years)
Time from Randomization or Treatment Initiation to Death due to any Cause for IMpower133 Participants Only | Day 1 (as indicated in parent study protocol) until death due to any cause (up to maximum 10 years or until the sponsor stop)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (170):
- United States (44):
  - HonorHealth Research Institute ? Bisgrove, Scottsdale, Arizona
  - Angeles Clinic & Rsch Inst, Los Angeles, California
  - UCLA, Los Angeles, California
  - Kaiser Permanente - San Diego (Zion Ave), San Marcos, California
  - University Of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Ctr - Denver (Williams), Denver, Colorado
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists - Fort Myers (Broadway), Fort Myers, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Florida Cancer Specialists., St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Inst., Tampa, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University Of Chicago Medical Center, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - New England Cancer Specialists, Westbrook, Maine
  - Johns Hopkins Univ Med Center, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Massachusetts General Hospital., Boston, Massachusetts
  - Beth Israel Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - US oncology research at Minnesota Oncology, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada - Eastern Avenue, Las Vegas, Nevada
  - Summit Medical Center, Florham Park, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Carolina BioOncology Institute, PLCC, Huntersville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oncology Associates of Oregon, P.C, Eugene, Oregon
  - Northwest Cancer Specialists - Portland (N Broadway), Portland, Oregon
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Res Inst, Nashville, Tennessee
  - Texas Oncology - DFW, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Fundación CENIT para la Investigación en Neurociencias, Buenos Aires, Argentina
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Princess AleXandra Hospital, Woolloongabba, Queensland
- Austria (2):
  - Klinik Penzing, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf, Vienna
- Belgium (2):
  - AZ Glorieux- vzw Werken Glorieux, Ronse
  - ZAS Sint Augustinus Wilrijk, Wilrijk
- Brazil (3):
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Fundacao Antonio Prudente, São Paulo, São Paulo
- Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia, Bulgaria
- Canada (7):
  - Royal Victoria Hospital, Barrie, Ontario
  - William Osler Health Centre, Brampton, Ontario
  - Lakeridge Health Corporation-Oshawa, Oshawa, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Cite de La Sante de Laval, Laval, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Bradford Hill Centro de Investigaciones Clinicas, Recoleta, Chile
- Czechia (2):
  - Masarykuv onkologicky ustav, Brno
  - Thomayerova nemocnice, Praha 4 - Krc
- France (14):
  - Hopital Jean Minjoz, Besançon
  - Chu Grenoble - Hopital Albert Michallon, Grenoble
  - Centre Leon Berard, Lyon
  - Hopital Nord, Marseille
  - Centre René Gauducheau - cancer Nantes - Atlantique, Nantes
  - Centre Antoine Lacassagne, Centre de Lutte Contre le Cancer (CLCC) de Nice, Nice
  - Hopital Saint Louis, Paris
  - GH Paris Saint Joseph, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CH de Saint Quentin, Saint-Quentin
  - Centre Medico-Chirurgical Foch, Suresnes
  - CHU de Toulouse - Hôpital Larrey, Toulouse
  - Institut Gustave Roussy, Villejuif
- Klinikum d.Universität München Campus Großhadern, München, Germany
- Hungary (2):
  - Semmelweis Egyetem X, Budapest
  - Református Pulmonológiai Centrum, Törökbálint
- Belinson Medical Center, Petah Tikva, Israel
- Italy (18):
  - Azienda Osp Uni Seconda Università Degli Studi Di Napoli, Napoli, Campania
  - Azienda Ospedaliera A. Cardarelli, Napoli, Campania
  - Istituto Nazionale per lo Studio e la Cura dei Tumori Fondazione G. Pascale, Napoli, Campania
  - A.O. Universitaria Policlinico Di Modena, Modena, Emilia-Romagna
  - Università Cattolica Del S Cuore, Rome, Lazio
  - IRCCS AOU San Martino - IST, Genoa, Liguria
  - ASL 3 Genovese, Genoa, Liguria
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO), Milan, Lombardy
  - Asst Di Monza, Monza, Lombardy
  - A.O.U. Maggiore della Carità, Novara, Piedmont
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano, Piedmont
  - Policlinico Vittorio Emanuele, Catania, Sicily
  - Azienda USL8 Arezzo-Presidio Ospedaliero 1 San Donato, Arezzo, Tuscany
  - A.O. Universitaria Pisana-Ospedale Cisanello, Pisa, Tuscany
  - Azienda Ospedaliera Universitaria Senese, U.O.C. Immunoterapia Oncologica, Siena, Tuscany
  - Ospedale Santa Maria Della, Perugia, Umbria
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
- Japan (8):
  - Shikoku Cancer Center, Ehime
  - Sendai Kousei Hospital, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Iwate Medical University Hospital, Numakunai
  - Okayama University Hospital, Okayama
  - Toranomon Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Respiratory Medicine, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- NKI/AvL, Amsterdam, Netherlands
- Auckland city hospital, Auckland, New Zealand
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Oddzia? Onkologii Klinicznej i Chemioterapii Szpitala ELBL?SKA, Warsaw
  - Narod.Inst.Onkol. im. M.Sklodowskiej - Curie-Panst.Inst.Bad, Warsaw
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar do Porto ? Hospital de Santo António, Porto
- Romania (2):
  - Institut Oncologic Ion Chiricuta, Cluj-Napoca
  - ONCOMED - Medical Centre, Timișoara
- Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast, Russia
- Serbia (2):
  - Clinic for Pulmonology, Clinical Center of Serbia, Belgrade
  - University Hospital Medical Center Bezanijska kosa, Belgrade
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Korea (4):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Samsung Medical Center, Seoul
- Spain (24):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Complejo Hospitalario Universitario A Coruña (CHUAC, Materno Infantil), Oncología, A Coruña, LA Coruna
  - Hospital Universitario Materno Infantil de Gran Canaria, Las Palmas de Gran Canaria, LAS Palmas
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clinic de Barcelona. Unidad de Nuevas Terapias, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital San Pedro De Alcantara, Cáceres
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital de Madrid Norte Sanchinarro- Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital NisA 9 de Octubre, Valencia
- CHUV, Lausanne, Switzerland
- Taiwan (3):
  - Changhua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - National Taiwan Uni Hospital, Taipei
- Thailand (3):
  - Chulalongkorn Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Faculty of Med. Siriraj Hosp., Bangkok
- Turkey (Türkiye) (3):
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital, Istanbul
  - Hacettepe Uni Medical Faculty Hospital, S?hhiye, Ankara
- Mun. Multifield Clin.Hosp.#4,Dept. of Chemotherapy, DSMU, Dnipropetrovsk, Ukraine
- United Kingdom (9):
  - Barts & London School of Med, London
  - Royal Free Hospital, London
  - St George's Hospital, London
  - Royal Marsden Hospital - London, London
  - Charing Cross Hospital, London
  - Christie Hospital NHS Trust, Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Nottingham City Hospital, Nottingham
  - Royal Marsden Hospital - Surrey, Surrey

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Reck M, Dziadziuszko R, Sugawara S, Kao S, Hochmair M, Huemer F, de Castro G Jr, Havel L, Bernabe Caro R, Losonczy G, Lee JS, Kowalski DM, Andric Z, Califano R, Veatch A, Gerstner G, Batus M, Morris S, Kaul M, Cuchelkar V, Li H, Danner BJ, Nabet BY, Liu SV. Five-year survival in patients with extensive-stage small cell lung cancer treated with atezolizumab in the Phase III IMpower133 study and the Phase III IMbrella A extension study. Lung Cancer. 2024 Oct;196:107924. doi: 10.1016/j.lungcan.2024.107924. Epub 2024 Aug 10. PMID 39306923